CLINICAL TRIAL: NCT07061665
Title: Cities for Better Health Childhood Obesity Prevention Initiative in JAPAN
Acronym: CBH COPI JAPAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiba University (Other)
Collaborators: Novo Nordisk A/S (Industry); The Behavioural Insights Team (Other); Delivery Associates (Unknown)
Responsible Party: Principal Investigator, Atsushi Nakagomi, Associate Professor, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M10825
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life (QOL); Nutrition; Physical Activity; Obesity; Childhood Obesity
Keywords: BMI; Childhood obesity; Japan; Chiba city; physical activity; nutrition; health equity; community intervention; randomized controlled trial; KIDSCREEN-10; Diet Quality Questionnaire
MeSH Terms: conditions — Motor Activity; Obesity; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This study employs a parallel interventional design. Participants, grouped by 22 school clusters (Junior High School Districts), are assigned to either an intervention group or a control group for the duration of the study. The intervention group receives a multi-level, multi-component program aimed at childhood obesity prevention, while the control group continues with usual practice. Data will be collected through repeated cross-sectional surveys at baseline, 1-year, and 2-year follow-up. Statistical analyses will use ANCOVA models, adjusted for baseline outcomes and clustering.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 11 Junior High School District (JHSD) clusters in Chiba City receive a multi-level, multi-component intervention targeting individual, environmental, and community factors for childhood obesity prevention.
  Interventions: Behavioral: Multi-level, Multi-component Intervention Package
- Control Group (No Intervention): 11 Junior High School District clusters in Chiba City serve as a comparator, continuing usual practices without new obesity prevention interventions from the study.

INTERVENTIONS:
Behavioral: Multi-level, Multi-component Intervention Package — The CBH COPI intervention applies multi-level strategies to improve children's environments and foster healthy behaviors. In schools, activities include schoolyard enhancements (e.g., hopscotch), inter-school sports events, nutrition lectures, healthy snacks, and educational materials linking health and academics. In parks and roads, improvements include cycling/walking promotions, signage, healthier vending machines, and community events. Supermarkets support healthy choices through menu information, loyalty incentives, cooking classes, product placement, and healthy food sales. At home and in communities, the Min-Challe app supports habit formation, with athletes, mascots, and ambassadors promoting healthy living. The coordinated program aims to naturally promote healthy eating, physical activity, and sustained lifestyle change among children aged 6-12 in Chiba City.
  Arms: Intervention Group

SUMMARY:
The goal of this interventional study is to prevent childhood obesity in children aged 6-12 years in Chiba City, Japan. The main questions it aims to answer are:

* Does the multi-component intervention for environments around children reduce the BMI z-score of children aged 6-12 years after one and two years?
* Does the multi-component intervention for environments around children improve the health-related quality of life (assessed by KIDSCREEN-10) of children aged 6-12 years after one and two years?

Researchers will compare school clusters receiving the intervention to control clusters to see if the intervention package promotes healthy eating, increases physical activity, improves health-related quality of life, and reduces obesity prevalence.

Participants will:

* Attend elementary schools within participating clusters (either the intervention or control group).
* Have baseline data collected, with follow-up assessments after one year and two years.
* Potentially participate in school-based programs (nutrition education, physical activity promotion) and community-based initiatives (park activation, supermarkets) if in an intervention cluster.
* Have their physical activity and dietary behavior assessed through self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years who are currently enrolled in one of the public elementary schools located within the 22 participating Junior High School District clusters in Chiba City.
* The parent or legal guardian of each child must provide written informed consent prior to participation.
* Parents or legal guardians must have sufficient Japanese language proficiency to understand study procedures, complete questionnaires, and provide accurate information during the study.
* Children must be physically and cognitively capable of participating in school- and community-based activities involved in the intervention.
* Participants must not have any medical conditions that would preclude safe participation in routine physical activities promoted by the intervention.

Exclusion Criteria:

* Children whose parents or legal guardians fail to provide complete informed consent.
* Families who withdraw consent at any point during the study period.
* Children who independently express refusal to participate, even with parental consent.
* Children with serious physical, psychological, or developmental disorders that prevent them from participating safely in the program's activities.
* Families planning to relocate outside of Chiba City during the study period, making follow-up assessment infeasible.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2200 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Body mass index z-score (BMI-z) adjusted for age and sex | Baseline, 1-year follow-up, 2-year follow-up (2025-2027)
  The primary outcome is the BMI z-score, calculated using the WHO 2007 Growth Reference. This metric standardizes a child's relative weight status by adjusting for both age and sex, enabling comparisons across different age groups and sexes. It represents the number of standard deviations a child's BMI is from the mean BMI of a healthy reference population. The BMI z-score allows for monitoring obesity-related changes over time and assessing the intervention's effectiveness in preventing excessive weight gain. The use of this z-score ensures consistency with international standards, facilitating global comparison of childhood obesity trends. The analysis will focus on changes in BMI z-score from baseline to 1-year and 2-year follow-ups.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL) | Baseline, 1-year follow-up, 2-year follow-up (2025-2027)
  HRQoL will be assessed using the KIDSCREEN-10 index, a validated, self-reported measure capturing children's subjective well-being across physical, emotional, social, and school functioning. This 11-item scale uses a 5-point Likert response for each item, which is then converted into a standardized T-score, further transformed to a 0-100 scale. On this scale, higher scores indicate better perceived quality of life. Changes in KIDSCREEN-10 scores will be tracked from baseline through 1-year and 2-year follow-ups to evaluate the intervention's impact on children's overall well-being.

OTHER OUTCOMES:
Physical Activity | Baseline, 1-year follow-up, 2-year follow-up (2025-2027)
  Physical activity will be assessed using self-reported daily minutes of moderate-to-vigorous physical activity (MVPA) and sedentary screen time. Participants will report time spent in activities such as sports, cycling, or active play, as well as screen-based sedentary behaviors. Data will be collected at baseline, 1-year, and 2-year follow-ups to evaluate the intervention's impact on physical activity patterns and sustained behavioral changes. Interpretation will be guided by international guidelines on daily activity targets.
Diet | Baseline, 1-year follow-up, 2-year follow-up
  Dietary outcomes will be assessed using the adapted Diet Quality Questionnaire (DQQ). This questionnaire evaluates children's usual intake of key food groups and dietary patterns. Participants or guardians will report the frequency of consuming various categories, including fruits, vegetables, whole grains, protein sources, dairy products, snacks, and sugary drinks. The DQQ aligns with global dietary guidelines and calculates scores reflecting dietary diversity and balance. Data will be collected at baseline, 1-year, and 2-year follow-ups to assess changes in dietary habits and the intervention's effects on promoting healthier eating patterns.

CONTACTS AND LOCATIONS:
Locations (1):
- Chiba University, Chiba, Chiba, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be shared with global collaborators (Novo Nordisk A/S, The Behavioural Insights Team, Oxford University) for pooled global analyses.
Supporting Information: Study Protocol